CLINICAL TRIAL: NCT03571841
Title: Sexual Health and Rehabilitation After Ovarian Suppression Treatment (SHARE-OS): An Educational Intervention for Young Breast Cancer Survivors
Brief Title: Sexual Health and Rehabilitation After Ovarian Suppression Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Howard Cox Fund for Women Assistant Professors (Unknown)
Responsible Party: Principal Investigator, Sharon Bober, Ph.D, Prinicipal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 18-140
Record Dates: First submitted 2018-06-18; First posted 2018-06-28 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Breast Cancer Survivors; Sexual Function Disturbances; Ovarian Suppression Treatment
Keywords: Breast Cancer Survivors; Sexual Function Disturbances; Ovarian Suppression Treatment
MeSH Terms: conditions — Sexual Dysfunctions, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Educational Intervention (Experimental): For breast cancer survivors currently on chemical ovarian suppression who are experiencing sexual dysfunction.
  * Group Session
  * Telephone Booster Session
  Interventions: Behavioral: Group Session; Behavioral: Telephone Booster

INTERVENTIONS:
Behavioral: Group Session — The 4-hour group session will be structured around three 60-minute modules and creation of a personal action plan
Behavioral: Telephone Booster — One month following the group session, women will receive a telephone booster session (<15 minutes). This brief telephone check-in is intended to help women review progress with their individualized action-plan, problem-solve around continuing problems, and plan for maintenance moving forward.

SUMMARY:
This research study is evaluating an educational intervention for breast cancer survivors who have experienced changes in sexual function after ovarian suppression treatment to reduce the risk of breast cancer recurrence.

DETAILED DESCRIPTION:
The purpose of this research is to study the effectiveness of an educational intervention for breast cancer survivors who have experienced changes in sexual function after ovarian suppression treatment to reduce the risk of cancer recurrence. The aim is to develop an effective intervention to help women manage these changes and restore sexual health and functioning.

- This study consists of attending a group educational session followed by a one-on-one telephone coaching session.

* The group educational session will last about 4 hours, and will include information on resources, self-help strategies, and relaxation techniques.
* The telephone coaching session will take place four weeks after the group session, and will last about 15 minutes

ELIGIBILITY:
Inclusion Criteria:

* Women with a history of breast cancer who are currently on chemical ovarian suppression
* Current age ≤ 50
* No active cancer therapy in the past 6 months and no future therapy planned
* Endorsement of at least one sexual symptom (see Appendix A for eligibility screening)
* English-speaking

Exclusion Criteria:

* History of pelvic radiation
* Prior participation in one of Dr. Bober's sexual health workshops

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Change in Sexual Function (FSFI) | Paired t-test (Wilcoxon signed-rank test) Baseline to 2 Month Follow-up
  Baseline to 2 Month Follow-up Paired t-test (Wilcoxon signed-rank test)

SECONDARY OUTCOMES:
Change in participants psychological distress on Brief Symptom Inventory | Baseline to 2 Months
  Paired t-test (Wilcoxon signed-rank test)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Bober, Ph.D, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States